CLINICAL TRIAL: NCT00467974
Title: A Randomized Controlled Trial of Transarterial Ethanol Ablation (TEA) With Lipiodol-Ethanol Mixture (LEM) Versus Transcatheter Arterial Chemoembolisation (TACE) for Unresectable Hepatocellular Carcinoma
Brief Title: Transarterial Ethanol Ablation (TEA) Versus Transcatheter Arterial Chemoembolisation (TACE) for Hepatocellular Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Edwin P Hui, Consultant, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC017
Record Dates: First submitted 2007-04-30; First posted 2007-05-01 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2014-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Tea; leukocyte endogenous mediator

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): TEA with LEM
  Interventions: Procedure: TEA with LEM
- 2 (Active Comparator): TACE
  Interventions: Procedure: TACE

INTERVENTIONS:
Procedure: TEA with LEM — Transarterial ethanol ablation (TEA) with Lipiodol-ethanol mixture (LEM)
  Arms: 1
Procedure: TACE — Transarterial chemoembolisation (TACE)
  Arms: 2

SUMMARY:
The current randomized controlled trial comparing LEM and TACE aims to evaluate the safety and efficacy of LEM as compared to TACE for treating patients with unresectable HCC.

DETAILED DESCRIPTION:
The standard loco-regional treatment for unresectable hepatocellular carcinoma is transarterial chemoembolization (TACE). However, The drawback of conventional chemoembolization (TACE) for liver cancer is that it cannot effectively embolize portal venules supplying the tumors, therefore chemoembolization is difficult to completely eradicate the tumor. Usually multiple treatments are required and tumor recurrences are common.

Transarterial Ethanol Ablation (LEM) can potentially provide a better treatment outcome with fewer treatment sessions. Preliminary results from a clinical study showed that the complication rate is reduced while survival rate may be improved. This study aims to compare survival duration and response rate between the treatments TACE and LEM.

ELIGIBILITY:
Inclusion Criteria:

Patient factor

* Age > 18
* Child-Pugh A or B cirrhosis
* ECOG performance status Grade 2 or below
* No serious concurrent medical illness
* No prior treatment (including surgery) for HCC

Tumor factor

* Histologically or cytologically proven HCC (an alphafetoprotein level > 500 ug/ml in the presence of radiological findings suggestive of HCC in a patient with chronic HBV or HCV infection can be considered eligible at investigator's discretion)
* Unresectable and locally advanced disease without extra-hepatic disease
* Massive expansive or nodular tumor morphology with measurable lesion on CT
* Size of largest tumor <= 15cm in largest dimension
* Number of main tumor <= 5, excluding associated small satellite lesions.

Exclusion Criteria:

Patient factor

* History of prior malignancy except skin cancer
* History of significant concurrent medical illness such as ischemic heart disease or heart failure
* History of acute tumor rupture
* Serum creatinine level > 180 umol/L
* Presence of biliary obstruction not amenable to percutaneous drainage
* Child-Pugh C cirrhosis

Evidence of poor liver function

* History of hepatic encephalopathy, or
* Intractable ascites not controllable by medical therapy, or
* History of variceal bleeding within last 3 months, or
* Serum total bilirubin level > 50 umol/L, or
* Serum albumin level < 28g/L, or
* INR > 1.3

Tumor factor

* Presence of extrahepatic metastasis
* Predominantly infiltrative lesion
* Diffuse tumor morphology with extensive lesions involving both lobes.

Vascular complications

* Hepatic artery thrombosis, or
* Partial or complete thrombosis of the main portal vein, or
* Tumor invasion of portal branch of contralateral lobe, or
* Hepatic vein tumor thrombus, or
* Significant arterioportal shunt not amenable to shunt blockage, or
* Significant arteriovenous shunt not amenable to shunt blockage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2007-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
overall survival | 3 years
progression free survival | 3 years

SECONDARY OUTCOMES:
tumor response | 4 weeks after end of treatment
rate of conversion to resectable stage | 4 weeks after end of treatment
toxicity of treatment | 4 weeks after end of treatment
quality of life | up to one year after randomisation
consumption of hospital resources | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Simon CH Yu, MD, FRCR, Principal Investigator — Department of Diagnostic Radiology and Organ Imaging, Prince of Wales Hospital, The Chinese University of Hong Kong
Locations (3):
- Hong Kong (3):
  - Department of Clinical Oncology, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong
  - Department of Diagnostic Radiology and Organ Imaging, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong
  - Department of Surgery, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong

REFERENCES:
- [Derived] Yu SC, Hui JW, Hui EP, Chan SL, Lee KF, Mo F, Wong J, Ma B, Lai P, Mok T, Yeo W. Unresectable hepatocellular carcinoma: randomized controlled trial of transarterial ethanol ablation versus transcatheter arterial chemoembolization. Radiology. 2014 Feb;270(2):607-20. doi: 10.1148/radiol.13130498. Epub 2013 Oct 28. PMID 24126369